CLINICAL TRIAL: NCT00415792
Title: Administration of Human Chorionic Gonadotropin (hCG) Versus Gonadotropin Releasing Hormone (GnRH) Agonist for Ovulation Induction in Hyper-Responder Patients
Brief Title: Comparison Between hCG and GnRH Agonist for Ovulation Induction in Patients With High Response to IVF Drugs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Eugonia (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: arvekap vs pregnyl
Record Dates: First submitted 2006-12-22; First posted 2006-12-25 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Infertility
Keywords: Ovulation induction; hCG; GnRH agonist; hyper-responders
MeSH Terms: conditions — Infertility | interventions — Chorionic Gonadotropin

INTERVENTIONS:
Drug: Arvekap, Pregnyl

SUMMARY:
hCG and GnRH agonist can be used to induce final oocyte maturation and ovulation in IVF cycles. These two approaches will be compared in this study in terms of pregnancy rates and embryological data using patients with hyper-response to IVF drugs.

DETAILED DESCRIPTION:
hCG is commonly used for the substitution of the endogenous LH surge to induce oocyte maturation and ovulation induction in ovarian hyperstimulation protocols for in vitro fertilization (IVF). However, hCG is related to the occurrence of the ovarian hyperstimulation syndrome (OHSS), a potentially life-threatening complication and hyper-responding patients are particularly in high risk. An alternative to exogenous hCG is the administration of a GnRH agonist inducing an endogenous rise in both LH and FSH levels due to the initial flare effect.

Comparisons: Pregnancy rates and embryological data will be compared from hyper-responding patients receiving either GnRH agonist (Arvekap) or hCG (Pregnyl) for ovulatrion induction following a GnRH antagonist treatment cycle.

ELIGIBILITY:
Inclusion Criteria:

* Hyper-responder patients (>20 oocytes retrieved)

Exclusion Criteria:

* Normal responders
* Poor responders
* PCOS

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2003-11; Study Completion 2005-07

PRIMARY OUTCOMES:
Ongoing pregnancy per embryo transfer

SECONDARY OUTCOMES:
Biochemical pregnancy per embryo transfer
Clinical pregnancy per embryo transfer
Embryological data

CONTACTS AND LOCATIONS:
Overall Officials: Tryfon Lainas, PhD, Principal Investigator — Eugonia
Locations (1):
- Eugonia, Athens, Greece

REFERENCES:
- [Background] Griesinger G, Diedrich K, Devroey P, Kolibianakis EM. GnRH agonist for triggering final oocyte maturation in the GnRH antagonist ovarian hyperstimulation protocol: a systematic review and meta-analysis. Hum Reprod Update. 2006 Mar-Apr;12(2):159-68. doi: 10.1093/humupd/dmi045. Epub 2005 Oct 27. PMID 16254001